CLINICAL TRIAL: NCT02028858
Title: Cannabis and Parkinson's Disease Tremor: A Natural History Study
Status: Completed | Type: Observational
Sponsor: Bastyr University (Other)
Responsible Party: Sponsor
Other Study IDs: 13A-1339
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, observational study designed to describe the effects of Cannabis on Parkinson's Disease tremor.

DETAILED DESCRIPTION:
Ten individuals with Parkinson's disease (PD) and tremor who use Cannabis were observed for two weeks. Individuals were asked to keep a journal of Cannabis use (form, delivery method, amount) and wear an accelerometer on the wrist with the dominant tremor. Analyses will be performed to describe whether Cannabis use affects PD tremor following use.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease
* Presence of PD-related tremor
* Currently using Cannabis for management of tremor
* Obtaining Cannabis in accordance with Washington State law
* Willing to log activities and experiences
* Willing to wear a motion sensor
* Able to attend 2 on-site visits

Exclusion Criteria:

* Presence of active infection within 5 days prior to enrollment
* Presence of unusual stressor within 5 days prior to enrollment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics; Washington State Parkinson's Disease Registry
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percent reduction in tremor as measured by Opal movement sensor | Upon enrollment, ongoing for 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K Mischley, ND, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States

IPD SHARING:
Plan to Share IPD: No